CLINICAL TRIAL: NCT05135871
Title: An Open-Label, Parallel-Group, Single-Center Phase 1 Clinical Study to Evaluate the Pharmacokinetics of a Single Oral Dose of Mavacamten in Healthy Adult Chinese Subjects
Brief Title: Study Evaluating the Pharmacokinetics of Mavacamten in Healthy Adult Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB2001-101
Record Dates: First submitted 2021-10-28; First posted 2021-11-26 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-06

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Mavacamten
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: Mavacamten 15 mg (Experimental): Cohort 1: 15 mg capsules × 1 on Day 1
  Interventions: Drug: Mavacamten
- Cohort 2: Mavacamten 25 mg (Experimental): Cohort 2: 10 mg capsules x 1 and 15 mg capsules x 1 on Day 1
  Interventions: Drug: Mavacamten
- Cohort 3: Mavacamten 15 mg (Experimental): Cohort 3: 15 mg capsules × 1 on Day 1
  Interventions: Drug: Mavacamten
- Cohort 4: Mavacamten 15 mg (Experimental): Cohort 4: 15 mg capsules × 1 on Day 1
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Single fasted oral dose of Mavacamten 15/25 mg on Day 1
  Other Names: Mavacamten capsule

SUMMARY:
Mavacamten is a small-molecule allosteric inhibitor of cardiac myosin that reversibly inhibits its binding to cardiac actin, thereby relieving systolic hypercontractility and improving ventricular compliance. This is an open-label, parallel-group, single-center Phase 1 clinical study. Healthy adult Chinese subjects with different genotypes will be included and administered with a single fasted oral dose of mavacamten to evaluate its PK profile. Up to 44 subjects will be enrolled in this study.

DETAILED DESCRIPTION:
Approximately 44 healthy adult Chinese subjects are expected to be enrolled in this study according to their genotypes into 4 cohorts.

The doses administered include: 15 mg for cohort 1; 25 mg for Cohort 2; 15 mg for Cohort 3; 15 mg for Cohort 4. Blood samples will be collected from subjects at scheduled time points for PK testing. Series of safety assessments (including but not limited to AEs, laboratory tests, vital signs, and ECGs) will be performed during the whole study at specified time points.

This study will consist of the following 5 periods:

* Pre-screening period and Screening period (Day -43 to Day -2, up to 42 days)
* In-house period (Day -1 to Day 3, total 4 days)
* Outpatient period (Day 4 to Day 75, total 72 days):
* End of study visit (Day 75)

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between the ages of 18 and 60 (inclusive) at screening
* With a body mass index (BMI) between 18 kg/m2 and 30 kg/m2 (inclusive) at screening
* Healthy as determined at screening and on Day -1
* Female subjects shall not be pregnant or breastfeeding
* Male partners of female subjects must also adopt a contraceptive method from screening through 5 months after administration of the investigational drug
* Able to understand and comply with the study procedures, understand the risks involved in this study, and provide written informed consent according to local and institutional guidelines before screening procedure

Key Exclusion Criteria:

* History of clinically significant arrhythmia
* History of any type of malignant tumors within 5 years of the Screening Visit
* Positive serologic tests at screening for infections with human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) antibody or hepatitis B virus (HBV) surface antigen at screening
* The vital signs of screening period and Day -1 were unqualified
* Subjects who have taken prescription medications within 28 days prior to screening or within 5 times of T1/2 (if known), whichever is longer
* History or evidence of any other clinically significant abnormalities, conditions, or diseases that, in the opinion of the investigator, would pose a risk to the safety of the subject or interfere with study evaluation, procedures, or its completion
* Any condition or treatment for a condition that might interfere with the conduct of the trial or might, in the opinion of the investigator, put the subject at risk, including but not limited to, alcoholism, drug dependence or abuse, and psychiatric conditions, if he/she participates in this study
* Positive test for alcohol or drug abuse at screening and on Day -1
* Use of tobacco within 28 days prior to screening
* Hypersensitivity to mavacamten or any of the components of its formulation
* Prior exposure to mavacamten
* Unable to comply with the study restrictions/requirements, including the number of required visits to the clinical site
* Unsuitable to participate in the study as judged by the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Chen N, Hsu P, Sun J, Li W, Wang Q, Samira M, Wei Q, Yu J, Cao G, Yang H, Wang L, Wang J, Jin Y, Liu W, Wu J, He J, Lyu C, Zhang J. Pharmacokinetics and safety of mavacamten in healthy Chinese participants with different CYP2C19 phenotypes. Clin Transl Sci. 2024 Jul;17(7):e13877. doi: 10.1111/cts.13877. PMID 39014868

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: Mavacamten 25 mg: Cohort 2: 10 mg capsules x 1 and 15 mg capsules x 1 on Day 1
  Mavacamten: Single fasted oral dose of Mavacamten 25 mg on Day 1
- Cohort 1: Mavacamten 15 mg: Cohort 1: 15 mg capsules × 1 on Day 1
  Mavacamten: Single fasted oral dose of Mavacamten 15 mg on Day 1
- Cohort 3: Mavacamten 15 mg: Cohort 3: 15 mg capsules × 1 on Day 1
  Mavacamten: Single fasted oral dose of Mavacamten 15 mg on Day 1
- Cohort 4: Mavacamten 15 mg: Cohort 4: 15 mg capsules × 1 on Day 1
  Mavacamten: Single fasted oral dose of Mavacamten 15 mg on Day 1
Period: Overall Study
Arm/Group | Cohort 2: Mavacamten 25 mg | Cohort 1: Mavacamten 15 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Started | 13 | 12 | 12 | 8
Completed | 12 | 12 | 12 | 8
Not Completed | 1 | 0 | 0 | 0
Not completed — 1 subject withdrew from the study before administration of the IMP due to pre-dose abnormal ECG | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Mavacamten 25 mg: Cohort 2: 10 mg capsules x 1 and 15 mg capsules x 1 on Day 1
  Mavacamten: Single fasted oral dose of Mavacamten 25 mg on Day 1 13 subjects were assigned to Cohort 2 but 1 subject (Cohort 2) withdrew from the study before administration of the study drug due to pre-dose abnormal ECG and was excluded from the pharmacokinetic analysis set and safety analysis set.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 8 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (4.99) | 31.0 (7.12) | 28.9 (6.32) | 35.4 (4.31) | 30.1 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 11
  Male | 9 | 9 | 9 | 6 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 12 | 12 | 12 | 8 | 44
  Non-Chinese | 0 | 0 | 0 | 0 | 0
  Han | 12 | 12 | 12 | 8 | 44
  Non-Han | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 12 | 12 | 12 | 8 | 44
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.34 (2.444) | 23.82 (2.571) | 23.26 (2.434) | 23.04 (2.312) | 23.67 (2.421)
CYP2C19 genotype [Count of Participants; unit: Participants]
  Ultra-rapid metabolizer | 0 | 0 | 0 | 0 | 0
  Rapid metabolizer | 1 | 1 | 0 | 0 | 2
  Normal metabolizer | 11 | 11 | 0 | 0 | 22
  Intermediate metabolizer | 0 | 0 | 12 | 0 | 12
  Poor metabolizer | 0 | 0 | 0 | 8 | 8
Left ventricular ejection fraction(%) [Mean (Standard Deviation); unit: %] | 68.0 (5.03) | 66.9 (396) | 66.4 (3.99) | 64.0 (5.58) | 66.5 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) (0-last), AUC(0-inf)
Description: Determination of pharmacokinetics parameters as measured by area under curve AUC(0-last), AUC(0-inf)
Time Frame: Predose, Day 1, Day 7, Day 10, Day 14, Day 21, Day 28, Day 35, Day 45, Day 67 and Day 75 post-dose
Population: One subject (Cohort 3) was excluded from the pharmacokinetic analysis set due to a major protocol deviation (use of prohibited drug moderate-acting CYP2C19 inhibitor "Omeprazole") affecting the assessment of PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 11 | 8
h*ng/mL
  (AUC) (0-last) | 9956 (35.61) | 20040 (50.49) | 18270 (21.05) | 39980 (23.60)
  AUC(0-inf) | 10030 (35.44) | 20280 (52.47) | 18430 (21.18) | 45810 (25.51)

2. Primary Outcome: Maximum Concentration (Cmax)
Description: Determination of pharmacokinetics parameters as measured by maximum concentration (Cmax)
Time Frame: Predose, Day 1, Day 7, Day 10, Day 14, Day 21, Day 28, Day 35, Day 45, Day 67 and Day 75 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 11 | 8
ng/mL | 395.4 (39.95) | 571.8 (25.69) | 485.2 (34.96) | 435.7 (35.66)

3. Primary Outcome: Time to Maximum Concentration (Tmax)
Description: Determination of pharmacokinetics parameters as measured by time to maximum concentration (Tmax)
Time Frame: Predose, Day 1, Day 7, Day 10, Day 14, Day 21, Day 28, Day 35, Day 45, Day 67 and Day 75 post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 11 | 8
h | 0.88 [0.50 to 3.00] | 1.50 [0.50 to 4.00] | 0.75 [0.50 to 3.00] | 0.63 [0.33 to 1.00]

4. Primary Outcome: Elimination Half-life (T1⁄2)
Description: Determination of pharmacokinetics parameters as measured by elimination half-life (T1⁄2)
Time Frame: Predose, Day 1, Day 7, Day 10, Day 14, Day 21, Day 28, Day 35, Day 45, Day 67 and Day 75 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 11 | 8
h | 120.3 (23.44) | 143.6 (42.32) | 205.4 (22.31) | 572.0 (25.03)

5. Primary Outcome: Apparent Volume of Distribution (Vd/F)
Description: Determination of pharmacokinetics parameters as measured by apparent volume of distribution (Vd/F)
Time Frame: Predose, Day 1, Day 7, Day 10, Day 14, Day 21, Day 28, Day 35, Day 45, Day 67 and Day 75 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 11 | 8
mL | 259500 (29.93) | 255300 (16.60) | 241200 (23.13) | 270200 (26.95)

6. Primary Outcome: Apparent Clearance (CL/F)
Description: Determination of pharmacokinetics parameters as measured by apparent clearance (CL/F)
Time Frame: Predose, Day 1, Day 7, Day 10, Day 14, Day 21, Day 28, Day 35, Day 45, Day 67 and Day 75 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mL/h
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 11 | 8
mL/h | 1495 (35.44) | 1233 (52.47) | 814.0 (21.18) | 327.5 (25.51)

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety assessments will be performed by incidence of adverse events during the whole study at specified time points
Time Frame: Up to 75 days
Population: All 44 subjects included in the safety analysis set: cohort 1 12 subjects, cohort 2 12 subjects, cohort 3 12 subjects, cohort 4 8 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 12 | 8
Participants
  Number of subjects with at least 1 AE | 3 | 6 | 9 | 3
  Number of subjects with at least 1 TEAE | 3 | 6 | 9 | 3
  Worst severity of TEAE(Mild) | 3 | 6 | 8 | 3
  Worst severity of TEAE(Moderate) | 0 | 0 | 1 | 0
  Worst severity of TEAE(Severe) | 0 | 0 | 0 | 0
  Drug-related TEAEs | 0 | 1 | 0 | 1
  TESAE | 0 | 0 | 0 | 0
  TEAE leading to study discontinuation | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0
  AESI | 0 | 0 | 0 | 0

8. Secondary Outcome: Body Weight at Screening and EOS
Description: Safety assessments will be performed by vital signs during the whole study at screening, Day-1, Day 3 and at the EOS Visit. A complete physical examination includes assessments of general appearance, skin, head and neck, chest, abdomen, back, spine, extremity neurological, and mental systems. Brief physical examination means chest examinations.
  Height (cm) and body weight (kg) will be measured at screening, and BMI (kg/m2) will be calculated. Body weight (kg) will be measured at EOS. The mean weight and the standard deviation are analysis for different cohort.
Time Frame: Body weight (kg) will be measured at screening (baseline) and EOS(75 days).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 12 | 8
kg
  Change from Baseline | 0.80 (2.899) | 0.70 (1.738) | -0.36 (2.378) | 1.25 (2.184)
  Baseline | 69.41 (12.699) | 62.78 (8.458) | 65.89 (11.157) | 68.26 (11.147)
  Day 75 | 70.21 (13.088) | 63.48 (9.405) | 65.53 (10.929) | 69.51 (11.530)

9. Secondary Outcome: Physical Examination Findings
Description: Safety assessments will be performed by physical examination findings during the whole study at specified time points
Time Frame: Up to 75 days
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 12 | 8
participants
  Number of abnormal but not clinically significant comprehensive physical examinations in baseline | 5 | 2 | 4 | 2
  Number of abnormal but not clinically significant comprehensive physical examinations in Day 75 | 5 | 2 | 4 | 2
  The number of abnormal with clinically significant comprehensive physical examinations in Day 75 | 0 | 1 | 0 | 0

10. Secondary Outcome: Heart Rate at Baseline and Day 75
Description: Safety assessments will be performed by electrocardiogram (ECG) parameters findings during the whole study at specified time points
Time Frame: Up to 75 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 12 | 8
beats/min
  Heart Rate-Baseline | 63.3 (8.70) | 63.0 (10.44) | 63.3 (10.44) | 62.8 (9.27)
  Heart Rate-D75 | 64.8 (7.12) | 66.4 (7.88) | 67.5 (5.35) | 66.8 (7.17)

11. Secondary Outcome: Clinical Laboratory Tests Data
Description: Safety assessments will be performed by clinical laboratory tests data(including hematology and blood chemistry, coagulation and urinalysis parameters) during the whole study at specified time points
Time Frame: Up to 75 days
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
Number analyzed (Participants) | 12 | 12 | 12 | 8
participants
  Blood fibrinogen increased | 0 | 0 | 1 | 1
  White blood cell count decreased | 0 | 1 | 0 | 1
  Alanine aminotransferase increased | 0 | 0 | 1 | 0
  Neutrophil count increased | 0 | 0 | 1 | 0
  Neutrophil count decreased | 0 | 0 | 0 | 1
  Eosinophil percentage increased | 0 | 0 | 1 | 0
  Eosinophil count increased | 0 | 0 | 1 | 0
  Urobilinogen urine increased | 0 | 0 | 0 | 1
  White blood cell count increased | 0 | 1 | 0 | 0
  Hemoglobin decreased | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: The study took about 80 days to monitor the adverse event for each subject.
Description: Consistent with clinicaltrials.gov definitions.
Arm/Group | Cohort 1: Mavacamten 15 mg | Cohort 2: Mavacamten 25 mg | Cohort 3: Mavacamten 15 mg | Cohort 4: Mavacamten 15 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 3/12 | 6/12 | 9/12 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Mavacamten 15 mg (N=12) | Cohort 2: Mavacamten 25 mg (N=12) | Cohort 3: Mavacamten 15 mg (N=12) | Cohort 4: Mavacamten 15 mg (N=8)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophil percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There are no special limitations and caveats to this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT05135871/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT05135871/SAP_001.pdf